CLINICAL TRIAL: NCT04856813
Title: Effectiveness of Massage Therapy With Active Component and Therapeutic Exercise in Cervical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Achalandabaso (Other)
Responsible Party: Sponsor-Investigator, Alexander Achalandabaso, Physiotherapy doctor, University of Jaén
Organization: University of Jaén (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2020/5/055
Record Dates: First submitted 2021-04-06; First posted 2021-04-23 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Neck Pain; Chronic Pain
Keywords: neck pain; exercise; Endurance; Training; Intervention
MeSH Terms: conditions — Neck Pain; Chronic Pain; Motor Activity | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: blind
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active (Experimental): this is the group that does a treatment with active movement, a program of pain education and a program of home exercise.
  Interventions: Other: Manual therapy active
- non active (Active Comparator): this is the group that does a treatment without active movement, a program of pain education and a program of home exercise.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy active — massage or ischemic compression with active contraction, tha will be isometric or concentric.
  Arms: active
Other: Manual therapy — massage or isquemic compression without contraction
  Arms: non active

SUMMARY:
It is an interventional study that proves the eficacy of the manual therapy with active manual therapy and combined with exercise in cervical pain.

DETAILED DESCRIPTION:
The study will be divided in two different groups:

* A control group (group A) : they will receive a treatment with manual therapy and physical exercise.
* An experimental group (group B) : they will receive the previous treatment, but also the pacient's do active muscle active contraction.

The exercise is compound by a home program of several exercises with diferent difficulties.

The contraction will consist on a combination of concentric and isometric work. being the patient's pain threshold the one that will guide us to the choice of the predominance of concentric or isometric contraction . Both groups will be joined by a five-minute work on pain education.

ELIGIBILITY:
Inclusion Criteria:

* accept to participate in the study, through informed consent
* subjects with chronic nonspecific neck pain lasting equal to or more than 3 months

Exclusion Criteria:

* Present neck pain caused by serious pathology such as: inflammatory, congenital, infectious, metabolic and neoplastic diseases.
* Cervical pathology of traumatic origin with less than 6 months of evolution.
* Rheumatic diseases.
* Neck pain with neurological signs such as: radiculopathy and myelopathy.
* Previous surgery of the cervical spine.
* Pregnancy.
* Have received physiotherapeutic treatment in the cervical region during the month prior to the inclusion of the study.
* Have the intention of receiving other physiotherapeutic treatments different from the one proposed during the study period.
* Present serious mental disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
Change in Neck disability | Baseline, 1 month (primary timepoint) , 2 months and 5 months after intervention commencement.
  Using the Neck Disability Index (NDI). It is made up of 10 items and each item is scored on a 6-point Likert scale (0 to 5), leading to a total score ranging from 0 to 50 (0 to 4 = no disability; 5 to 14 = mild disability; 15 to 24 = moderate disability; 25 to 34 = severe disability; and 35 to 50 = complete disability).

SECONDARY OUTCOMES:
Change in pain perception | Baseline, 1 month (primary timepoint), 2 months and 5 months after intervention commencement.
  Using the Visual Analog Scale (VAS) from 0 to 10
Change in Range of motion (ROM) | Baseline, 1 month (primary timepoint) and 2 months after intervention commencement.
  Using a inclinometer
Change in craniocervical flexion | Baseline, 1 month (primary timepoint) and 2 months after intervention commencement.
  Using the craniocervical flexion test (CCFT) we make a evaluation of the strength of the deep cervical flexor muscles. From 22 to 30 mmHg of preasure.
Change in kinesophobia | Baseline, 1 month (primary timepoint) , 2 months and 5 months after intervention commencement.
  Using the Tampa Scale for Kinesiophobia-11 (TSK-11), self-report of 17 items that address fear of movement and injury relapse. Four of the items are negatively written and scored inverse (4, 8, 12 and 16). The scores are added together to obtain a total score, with higher values reflecting greater kinesiophobia.
Change in Catastrophism | Baseline, 1 month (primary timepoint), 2 months and 5 months after intervention commencement.
  Using the Pain catastrophizing scale from 0 to 56
Change in Sleep Quality | Baseline, 1 month (primary timepoint) , 2 months and 5 months after intervention commencement.
  Using the Pittsburgh Sleep Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, Study Director — University of Jaen
Locations (1):
- Alexander achalandabaso, Alcalá de Henares, Madrid, Spain